CLINICAL TRIAL: NCT01747148
Title: A Phase 1, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of AVI-7100 in Healthy Subjects
Brief Title: Testing the AVI-7100 Flu Drug in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: 130029; 13-I-0029
Record Dates: First submitted 2012-12-08; First posted 2012-12-11 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12-21

CONDITIONS: Influenza
Keywords: Antisense; Influenza; IV Injection; RNA Based Therapeutic; RNA Interference
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Drug: AVI-7100 versus placebo — dose-escalating AVI-7100 versus placebo

SUMMARY:
Background:

- Influenza (flu) is a virus that causes people to get sick. Most of the time, the flu causes only a mild illness, but some people can become seriously ill or even die from it. Currently, some pills and inhaled powders can be used to treat the flu, but they only make flu symptoms end about a day sooner. More treatment choices for the flu are needed, especially for those who become seriously ill. Researchers want to test a new drug, AVI-7100, that might keep a person who takes it from having a more serious case of the flu.

Objectives:

- To see how healthy adult volunteers tolerate the AVI-7100 anti-influenza drug.

Eligibility:

- Healthy volunteers of normal weight between 18 and 60 years of age.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. A heart function test will also be performed.
* Participants will have either AVI-7100 or a placebo infusion. They will not know which infusion they have. . Participants will stay at the clinical center for a total of 8 hours after the infusion. Blood samples will be collected 1, 2, 4, and 8 hours after the end of the infusion
* Participants will return on Days 1, 2, 4, 10, and 28 after receiving the drug. Blood and urine samples will be collected. A heart function test will also be performed.
* There will be a second part of the study that is separate from the first one. Additional people will receive either AVI-7100 or placebo to test their reactions to a specific dose.

DETAILED DESCRIPTION:
Despite currently available antivirals, influenza causes significant morbidity and mortality (estimated 36,000 deaths each year in the United States alone). More agents are needed in the armamentarium of anti-influenza medications including novel mechanisms of action and parenteral agents.

This study will evaluate the safety of a novel RNA based therapeutic AVI-7100. Beginning with a low single-dose, subjects are randomized to receive either AVI-7100 or placebo and evaluated on Study Days 0, 1, 2, 4, 10, 28. The safety and tolerability is evaluated using symptoms, clinical laboratory tests, ECG, and pharmacokinetics. Utilizing a series of stopping rules and a medical monitor, the dose will be escalated as safety and tolerability are established. Once the maximum tolerated dose (MTD) is established in the first part of this study (either limited by adverse effects or up to maximum anticipated dose), the safety and tolerability of multi-dose administration will begin (replicating anticipated clinical use). Subjects again are randomized to either AVI-7100 or placebo daily for 5 days, and evaluated on Study Days 0, 1, 2, 3, 4, 5, 6, 8, 14, and 32. The dose used in the multi-dose cohorts will also be escalated as safety and tolerability are established.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 18 years and less than or equal to 60 years
  2. Body mass index (BMI) of 19-32 kg/m(2)
  3. Estimated glomerular filtration rate greater than or equal to 90 mL/min at screening, calculated using the MDRD formula
  4. Subjects must agree to:
* Not take any prescription or OTC medications with the exception of Tylenol, vitamins, seasonal allergy medications, and/or contraceptive medications for a period 7 days prior and during study drug administration.
* Not consume any alcohol for a period 2 days prior to and during study drug administration.

  5. One of the following in order to avoid pregnancy:
* Females who are able to become pregnant (i.e., are not postmenopausal)
* have not undergone surgical sterilization, and are sexually active with men) must agree to use at least 2 effective forms of contraception.
* From the date of the subject s signing of the informed consent form through 28 days after the last dose of study drug. At least one of the methods of contraception should be a barrier method.
* Males who have not undergone surgical sterilization and are sexually active with women must agree to use condoms plus have a partner use at least one additional effective form of contraception from the date of the subject s signing of the informed consent form through 28 days after the last dose of study drug.

EXCLUSION CRITERIA:

1. Any chronic medical problem that requires daily oral medications (except Tylenol, oral contraceptives, vitamins, and seasonal allergy medications), or other medical history that in the opinion of the investigator significantly increases the risk associated with a phase I drug.
2. History of cardiovascular disease or unexplained syncope
3. Women who are breast-feeding.
4. Positive urine or serum pregnancy test.
5. Abnormal ECG

   -defined as any clinically significant baseline Grade 1 or greater toxicity, or any Grade 3 or greater toxicity (regardless of clinical significance) by the toxicity table.

   --evaluating PR interval, QTc interval and rhythm.
6. Abnormal chemistry panel

   -defined as any clinically significant baseline Grade 1 or greater toxicity, or any Grade 3 or greater toxicity (regardless of clinical significance) by the toxicity table

   --evaluating only sodium [Na], potassium [K], serum bicarbonate [total CO2], creatinine, glucose,albumin, ALT, AST, ALKP, GGT, total bilirubin, LDH, and estimated GFR by the MDRD equation.
7. Abnormal complete blood count (CBC)

   -defined as any clinically significant baseline Grade 1 or greater toxicity, or any Grade 3 or greater toxicity (regardless of clinical significance) by the toxicity table

   -- evaluating only the WBC (to include absolute neutrophil and lymphocyte counts), hemoglobin, hematocrit, and platelets.
8. Abnormal urinalysis

   -defined as any clinically significant baseline Grade 1 or greater toxicity

   --evaluating only protein, and RBCs.
9. Urine-albumin-to-creatinine ratio (UACR) >30 mg/g.
10. Positive serology for Hepatitis B surface antigen.
11. Positive serology for Hepatitis C.
12. Positive serology for HIV-1.
13. Positive urine drug screen.
14. Participation in a study with receipt of any investigational drug within 5 half-lives or 30 days, whichever is longer, prior to study drug administration (i.e., Day 0)
15. Donation of blood or blood products within 30 days or plasma within 2 weeks prior to study drug administration (i.e., Day 0)
16. Receipt of blood products within 2 months prior to study drug administration (i.e., Day 0)
17. Receipt of any vaccination within 30 days prior to study drug administration (i.e., Day 0)
18. Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject s ability to complete and/or participate in this clinical study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2012-12-08; Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of AVI-7100 in healthy adults, following single- or multiple-dose, intravenous administration at escalating dose-levels | 2 years

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of intravenously administered AVI-7100 in healthy adults, following single- or multiple-dose, intravenous administration at escalating dose-levels | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Davey, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Novel Swine-Origin Influenza A (H1N1) Virus Investigation Team; Dawood FS, Jain S, Finelli L, Shaw MW, Lindstrom S, Garten RJ, Gubareva LV, Xu X, Bridges CB, Uyeki TM. Emergence of a novel swine-origin influenza A (H1N1) virus in humans. N Engl J Med. 2009 Jun 18;360(25):2605-15. doi: 10.1056/NEJMoa0903810. Epub 2009 May 7. PMID 19423869
- [Background] Abe T, Mizuta T, Hatta T, Miyano-Kurosaki N, Fujiwara M, Takai K, Shigeta S, Yokota T, Takaku H. Antisense therapy of influenza. Eur J Pharm Sci. 2001 Apr;13(1):61-9. doi: 10.1016/s0928-0987(00)00208-6. PMID 11292569
- [Background] Mizuta T, Fujiwara M, Abe T, Miyano-Kurosaki N, Yokota T, Shigeta S, Takaku H. Inhibitory effects of an antisense oligonucleotide in an experimentally infected mouse model of influenza A virus. Biochem Biophys Res Commun. 2000 Dec 9;279(1):158-61. doi: 10.1006/bbrc.2000.3924. PMID 11112432
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-I-0029.html